CLINICAL TRIAL: NCT00376818
Title: Evaluation of a Stress Reduction Program in Patients With Malignant Brain Tumors and Their Family Caregivers
Brief Title: Stress Reduction Program in Patients With Malignant Brain Tumors and Their Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2306; P30CA043703 (NIH)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-06

CONDITIONS: Brain and Central Nervous System Tumors; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; adult medulloblastoma; adult anaplastic meningioma; adult papillary meningioma; adult mixed glioma; recurrent adult brain tumor; adult glioblastoma; adult grade III meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Medulloblastoma; Meningioma; Glioma; Brain Neoplasms | interventions — Yoga; Early Intervention, Educational; Surveys and Questionnaires; Mind-Body Therapies; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: exercise intervention — All participants will convene once per week for 8 weeks for a 90-minute session that will be based on yoga principles for a stress reduction.
  Other Names: Yoga
Other: educational intervention — A 15-minute educational session on a particular topic (mind-body connection; fight or flight response; relaxation response; the science and philosophy of yoga; the science of meditation; sleeping well; mindfulness; the healer within - how to harness your innate healing potential).
Other: physiologic testing — Both patients and family caregivers will complete Perceived Stress Scale (PSS) and Beck Anxiety Inventory (BAI) questionnaires.
  Other Names: questionnaire
Other: management of therapy complications — Brain Cancer module-20 questionnaire to assesses problems specific to brain tumor.
  Other Names: questionnaire
Behavioral: mind-body intervention procedure — Meditation practice in this study will consist of 15 minutes of "body scan" to completely relax the body from head to toe and will be followed by 15 minute silence during which the study participants will maintain awareness of their breath, bodily sensations and thoughts as they spontaneously arise. The remainder of the class will be devoted to a group discussion of personal reflections and challenges.
  Other Names: Meditation
Procedure: Measurement of stress-related hormones — Measurements of stress-related hormones: Stress hormones cortisol, dehydroepiandrosterone sulfate (DHEAS) and melatonin will be measured in saliva because their levels in saliva accurately reflect blood levels (Carlson et al, 2004). The non-invasive saliva collection method by cotton swabs (Salivette® by Sardstedt Inc.) will be used in this study.
  Other Names: salivary samples

SUMMARY:
RATIONALE: Yoga, meditation, and breathing exercises may help lower stress and improve quality of life in patients with malignant brain tumors and their family caregivers.

PURPOSE: This clinical trial is studying how well a stress reduction program works to improve the quality of life of patients with malignant brain tumors and their family caregivers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether regular practice of a stress reduction program for 8 weeks improves the quality of life of patients with malignant brain tumors.

Secondary

* Determine whether regular practice of a stress reduction routine decreases perception of stress and anxiety and stress- and inflammation-related hormones in both patients with malignant brain tumors and their primary family caregivers.

OUTLINE: This is a pilot study.

Patients and caregivers receive a 90-minute stress-reduction session once a week for 8 weeks. Each session comprises an educational session on stress reduction and yoga therapy comprising specific yoga postures, breathing exercises, and relaxation and meditation.

Quality of life, stress, anxiety, and levels of stress-related hormones (cortisol, dehydroepiandrosterone sulfate [DHEAS], and melatonin) are assessed at baseline and at week 8.

After completion of study treatment, patients and caregivers are followed at 6 and 12 months.

PROJECTED ACCRUAL: A total of 14 caregiver/patient pairs will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant brain tumor of 1 of the following subtypes:

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Astrocytoma WHO grade IV
  * Malignant meningioma
  * Anaplastic oligodendroglioma
  * Anaplastic oligoastrocytoma
  * Gliosarcoma
  * Anaplastic ependymoma
  * Medulloblastoma
* Caregivers must meet the following criteria:

  * Primary family caregiver
  * Age 18 and over

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%*
* Absolute neutrophil count ≥ 1,500/mm³*
* Platelet count ≥ 100,000/mm³*
* Bilirubin ≤ 2 times normal*
* Alkaline phosphatase ≤ 2 times normal*
* SGOT ≤ 3 times normal*
* BUN or creatinine ≤ 1.5 times normal*
* No other prior (within the past 3 years) or concurrent malignancies except for surgically cured carcinoma in situ of the cervix or nonmelanoma skin cancer*
* Not pregnant**
* Negative pregnancy test**
* Fertile patients must use effective contraception**
* No active infection**
* No medical condition that would interfere with the practice of yoga and meditation** NOTE: *Patient

NOTE: **Patient and caregiver

PRIOR CONCURRENT THERAPY:

* No other prior or concurrent stress reduction techniques using yoga or meditation*
* Concurrent standard or investigational chemotherapy, hormonal therapy, immunotherapy, biologic agents, or other complementary and alternative therapies as the primary or adjuvant treatment allowed (patient)
* No concurrent glucocorticoids (caregiver)
* Concurrent dexamethasone allowed provided the daily dose is < 2 mg/day (patient)
* No concurrent dehydroepiandrosterone sulfate (DHEAS) and/or melatonin supplements* NOTE: *Patient and caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Quality of life as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 Items (EORTC QLQ-C30) and Brain Cancer Module-20 | 12 months

SECONDARY OUTCOMES:
Decrease in perception of stress and anxiety in patients and their primary family caregivers as measured by the Perceived Stress Scale and Beck Anxiety Inventory questionnaires | 12 months
Decrease in stress- and inflammation-related hormones in patients and their primary family caregivers as measured by saliva samples | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Glen H. J. Stevens, DO, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States